CLINICAL TRIAL: NCT01776554
Title: A Phase II, Randomized, Observer-Blind, Multi-Center, Study to Evaluate Safety, Tolerability and Immunogenicity of an Adjuvanted Cell Culture-Derived H5N1 Subunit Influenza Virus Vaccine at Two Different Formulations in Healthy Pediatric Subjects.
Brief Title: Safety and Immunogenicity of Two Doses of H5N1 Influenza Vaccine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V89_11
Record Dates: First submitted 2013-01-20; First posted 2013-01-28 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Pandemic H5N1 Influenza
Keywords: Influenza, Pandemic, H5N1, Children
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- aH5N1c-High dose (Experimental)
  Interventions: Biological: Adjuvanted H5N1 pandemic influenza vaccine
- aH5N1c-Low dose (Experimental)
  Interventions: Biological: Adjuvanted H5N1 pandemic influenza vaccine

INTERVENTIONS:
Biological: Adjuvanted H5N1 pandemic influenza vaccine — Comparison of two doses of aH5N1c vaccine

SUMMARY:
Evaluate Safety, Tolerability and Immune response of adjuvanted H5N1 cell culture derived influenza vaccine in children.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pediatric subjects 6 months to 17 years of age,
2. Individuals' parent(s) or legal guardian(s) willing to provide written informed consent,
3. Individuals in good health,
4. Individuals/Individuals' parent(s)/legal guardian(s) willing to allow for serum samples to be stored beyond the study period,
5. Individuals willing to provide informed assent (where applicable).

Exclusion Criteria:

1. Individuals' parent(s)/legal guardian(s) not able to understand and follow study procedures,
2. History of any significant illness,
3. History of any chronic medical condition or progressive disease,
4. Presence of medically significant cancer,
5. Known or suspected impairment/alteration of immune function,
6. Presence of any progressive or severe neurologic disorder,
7. Presence of any bleeding disorders or conditions that prolongs bleeding time,
8. History of allergy to vaccine components,
9. Receipt of any other investigational product within 30 days prior to entry into the study,
10. History of previous H5N1 vaccination,
11. Receipt of any other type of seasonal vaccination within 2 months prior to entry into the study,
12. Receipt of any other vaccine within 2 weeks prior to entry into the study,
13. Body temperature ≥38°C (≥100.4° F) and/or acute illness within 3 days of intended study vaccination,
14. Pregnant or breast feeding,
15. Females of childbearing potential refusing to use acceptable method of birth control,
16. Body mass index (BMI) ≥ 35 kg/m2,
17. History of drug or alcohol abuse,
18. Any planned surgery during study period,
19. Individuals conducting the study and their immediate family members,
20. Individuals with behavioral or cognitive impairment or psychiatric diseases,
21. Individuals diagnosed with any growth disorders.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 662 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (12):
- United States (10):
  - 3 Meridian Clinical Research, Miami, Florida
  - 7 Heartland Research Associates, Newton, Kansas
  - 5 Heartland Research Associates, Wichita, Kansas
  - 9 Heartland Research Associates, Wichita, Kansas
  - 1 Saint Louis University, St Louis, Missouri
  - 6 Meridian Clinical Research, Omaha, Nebraska
  - 10 Tekton Research, Georgetown, Texas
  - 8 Foothill Family Clinic, Salt Lake City, Utah
  - 4 Foothill Family Clinic, South Cottonwood Heights, Utah
  - 2 Rockwood Clinic P S, Spokane, Washington
- Thailand (2):
  - 75 Phramongkutklao Hospital, Bangkok
  - 76 Faculty of Tropical Medicine Mahidol University, Bangkok

REFERENCES:
- [Derived] Chanthavanich P, Versage E, Van Twuijver E, Hohenboken M. Antibody responses against heterologous A/H5N1 strains for an MF59-adjuvanted cell culture-derived A/H5N1 (aH5N1c) influenza vaccine in healthy pediatric subjects. Vaccine. 2021 Nov 16;39(47):6930-6935. doi: 10.1016/j.vaccine.2021.10.010. Epub 2021 Oct 25. PMID 34711436
- [Derived] Chanthavanich P, Anderson E, Kerdpanich P, Bulitta M, Kanesa-Thasan N, Hohenboken M. Safety, Tolerability and Immunogenicity of an MF59-adjuvanted, Cell Culture-derived, A/H5N1, Subunit Influenza Virus Vaccine: Results From a Dose-finding Clinical Trial in Healthy Pediatric Subjects. Pediatr Infect Dis J. 2019 Jul;38(7):757-764. doi: 10.1097/INF.0000000000002345. PMID 31194712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 10 centers in United States and 2 centers in Thailand.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- High Dose: Subjects received 2 injections of a high dose of cell culture-derived adjuvanted monovalent inactivated subunit H5N1 vaccine three weeks apart.
- Low Dose: Subjects received 2 injections of a low dose of cell culture-derived adjuvanted monovalent inactivated subunit H5N1 vaccine three weeks apart.
Period: Overall Study
Arm/Group | High Dose | Low Dose
Started | 332 | 330
Completed | 315 | 307
Not Completed | 17 | 23
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Lost to Follow-up | 6 | 9
Not completed — Administrative Reason | 2 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Unclassified | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Low Dose | Total
Number analyzed (Participants) | 332 | 330 | 662
Age, Continuous [Mean (Standard Deviation); unit: Months] | 78.7 (55.9) | 78.1 (55.6) | 78.4 (55.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 152 | 164 | 316
  MALE | 180 | 166 | 346

OUTCOME MEASURES:

1. Primary Outcome: The Percentages Of Subjects Aged 6 to <36 Months, Achieving Hemagglutination Inhibition (HI) Titers ≥40 Against A/H5N1 Strain
Description: The optimal aH5N1c vaccine formulation was evaluated in terms of percentages of subjects aged 6 to <36 months, achieving HI titers ≥40 against homologous A/H5N1 strain, three weeks after second vaccination with either low dose or high dose of aH5N1c vaccine, according to the Center for Biologics Evaluation and Research (CBER) criterion.
  As there is no CBER criteria defined for children, immunogenicity was evaluated using CBER criterion applicable for adults (18-64 years).
  CBER criterion is met if the lower limit of the two-sided 95% confidence interval (CI) for the percentages of subjects achieving HI titer ≥40 meets or exceeds 70%.
Time Frame: Three weeks after 2nd vaccination (day 43)
Population: Analysis was done on the Full Analysis Set (FAS) i.e., the subjects who actually received at least one dose of study vaccination and provided at least one evaluable serum sample both before (baseline) and after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 93 | 90
Percentages of subjects
  Day 1 | 1 [0.027 to 6] | 0 [0 to 4]
  Day 43 (N=91,85) | 98 [92 to 100] | 94 [87 to 98]

2. Primary Outcome: The Percentages Of Subjects Aged 3 to <9 Years, Achieving HI Titers ≥40 Against A/H5N1 Strain
Description: The optimal aH5N1c vaccine formulation was evaluated in terms of percentages of subjects aged 3 to <9 years, achieving HI titers ≥40 against homologous A/H5N1 strain, three weeks after second vaccination with either low dose or high dose of aH5N1c vaccine, according to the CBER criterion.
  As there is no CBER criteria defined for children, immunogenicity was evaluated using CBER criterion applicable for adults (18-64 years).
  CBER criterion is met if the lower limit of the two-sided 95% CI for the percentages of subjects achieving HI titer ≥40 meets or exceeds 70%.
Time Frame: Three weeks after 2nd vaccination (day 43)
Population: Analysis was done on FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 98 | 101
Percentages of subjects
  Day 1 | 0 [0 to 4] | 0 [0 to 4]
  Day 43 (N=94,98) | 98 [93 to 100] | 86 [77 to 92]

3. Primary Outcome: The Percentages Of Subjects Aged 9 to <18 Years, Achieving HI Titers ≥40 Against A/H5N1 Strain
Description: The optimal aH5N1c vaccine formulation was evaluated in terms of percentages of subjects aged 9 to <18 years, achieving HI titers ≥40 against homologous A/H5N1 strain, three weeks after second vaccination with either low dose or high dose of aH5N1c vaccine, according to the CBER criterion.
  As there is no CBER criteria defined for children, immunogenicity was evaluated using CBER criterion applicable for adults (18-64 years).
  CBER criterion is met if the lower limit of the two-sided 95% CI for the percentages of subjects achieving HI titer ≥40 meets or exceeds 70%.
Time Frame: Three weeks after 2nd vaccination (day 43)
Population: Analysis was done on FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 103 | 109
Percentages of subjects
  Day 1 | 2 [0 to 7] | 1 [0.023 to 5]
  Day 43 (N=102,105) | 92 [85 to 97] | 79 [70 to 86]

4. Primary Outcome: The Percentages Of Subjects Aged 6 to <36 Months, Achieving Seroconversion Against A/H5N1 Strain
Description: Immunogenicity was measured in terms of the percentages of subjects aged 6 to <36 months, achieving seroconversion or significant increase in HI titer against the vaccine strain, three weeks after receiving two injections of low dose or high dose of aH5N1c vaccine according to the CBER criteria.
  Seroconversion is defined as the percentages of subjects with a prevaccination HI titer <10, a postvaccination titer ≥40; or in subjects with prevaccination HI titer ≥10, and a minimum four-fold rise in postvaccination HI antibody titer.
  CBER criterion is met if the lower limit of the two-sided 95% CI for the percentages of subjects achieving seroconversion for HI antibody titer meets or exceeds 40%.
Time Frame: Three weeks after 2nd vaccination (day 43)
Population: Analysis was done was FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 84 | 85
Percentages of subjects | 99 [94 to 100] | 94 [87 to 98]

5. Primary Outcome: The Percentages Of Subjects Aged 3 to <9 Years, Achieving Seroconversion Against A/H5N1 Strain
Description: Immunogenicity was measured in terms of the percentages of subjects aged 3 to <9 years, achieving seroconversion or significant increase in HI titer against the vaccine strain, three weeks after receiving two injections of low dose or high dose of aH5N1c vaccine according to the CBER criteria.
  Seroconversion is defined as the percentages of subjects with a prevaccination HI titer <10, a postvaccination titer ≥40; or subjects with prevaccination HI titer ≥10, and a minimum four-fold rise in postvaccination HI antibody titer.
  CBER criterion is met if the lower limit of the two-sided 95% CI for the percentages of subjects achieving seroconversion for HI antibody titer meets or exceeds 40%.
Time Frame: Three weeks after 2nd vaccination (day 43)
Population: Analysis was done on FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 93 | 98
Percentages of subjects | 98 [92 to 100] | 86 [77 to 92]

6. Primary Outcome: The Percentages Of Subjects Aged 9 to <18 Years, Achieving Seroconversion Against A/H5N1 Strain
Description: Immunogenicity was measured in terms of the percentages of subjects aged 9 to <18 years, achieving seroconversion or significant increase in HI titer against the vaccine strain, three weeks after receiving two injections of low dose or high dose of aH5N1c vaccine according to the CBER criteria.
  Seroconversion is defined as the percentages of subjects with a prevaccination HI titer <10, a postvaccination titer ≥40; or in subjects with prevaccination HI titer ≥10, and a minimum four-fold rise in postvaccination HI antibody titer.
  CBER criterion is met if the lower limit of the two-sided 95% CI for the percentages of subjects achieving seroconversion for HI antibody titer meets or exceeds 40%.
Time Frame: Three weeks after 2nd vaccination (day 43)
Population: This analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 102 | 105
Percentages of subjects | 92 [85 to 97] | 79 [70 to 86]

7. Primary Outcome: Number of Subjects (6 Month - <6 Years) Reporting Solicited Local and Systemic Adverse Events, After Any Vaccination
Description: Safety was assessed using the number of subjects who reported solicited local and systemic adverse events following vaccination with either low or high dose of aH5N1c vaccine.
Time Frame: From day 1 through day 7 after each vaccination.
Population: Analysis was done on the safety dataset, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Number of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 166 | 164
Number of subjects
  Any Local | 89 | 92
  Injection site erythema (N=159,162) | 4 | 2
  Injection site induration (N=159,162) | 2 | 2
  Injection site ecchymosis (N=159,162) | 0 | 1
  Injection site tenderness (N=159,162) | 89 | 91
  Any Systemic | 68 | 65
  Change in eating habits (N=159,162) | 29 | 20
  Irritability (N=159,162) | 47 | 45
  Sleepiness (N=159,162) | 40 | 40
  Fever (≥38°C; N=160,162) | 25 | 13
  Prevention of pain and/or fever (N=160,161) | 18 | 25
  Treatment of pain and/or fever (N=160,161) | 37 | 26
  Fever (≥40°C; N=160,162) | 1 | 0

8. Primary Outcome: Number of Subjects (≥6 Years - 17 Years) Reporting Solicited Local and Systemic Adverse Events, After Any Vaccination
Description: as for outcome 7
Time Frame: From day 1 through day 7 after any vaccination.
Population: Analysis was done on the safety dataset.
Measure: Number; unit: Number of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 163 | 165
Number of subjects
  Any Local | 111 | 115
  Injection site erythema (N=163,161) | 2 | 0
  Injection site induration (N=163,160) | 4 | 2
  Injection site ecchymosis (N=163,160) | 0 | 0
  Injection site pain (N=163,160) | 111 | 115
  Any Systemic | 79 | 82
  Myalgia (N=162,160) | 49 | 44
  Arthralgia (N=162,160) | 21 | 19
  Headache (N=162,160) | 36 | 47
  Fatigue (N=162,160) | 43 | 48
  Loss of Appetite (N=162,160) | 22 | 18
  Malaise (N=162,160) | 40 | 38
  Fever (≥38°C; N=163,161) | 7 | 5
  Prevention of pain and/or fever (N=163,161) | 14 | 10
  Treatment of pain and/or fever (N=163,161) | 24 | 23
  Fever (≥40°C; N=163,161) | 0 | 0
  Nausea (N=162,160) | 21 | 26

9. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Any Vaccination
Description: Safety was assessed using the number of subjects who reported any unsolicited adverse events, adverse events possibly or probably related to study vaccine, serious adverse events (SAEs), new onset of chronic diseases (NOCDs), medically attended AEs, AEs of special interest (AESIs), AEs leading to withdrawal from study following vaccination with either low or high dose of aH5N1c vaccine.
Time Frame: Any unsolicited AEs - day 1 through day 22 after any vaccination; SAEs, NOCDs. medically attended AEs, AESIs, AEs leading to study withdrawal- day 1 to day 387
Population: Analysis was done on the safety dataset.
Measure: Number; unit: Number of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 329 | 329
Number of subjects
  Any AEs | 149 | 156
  At least possibly related AEs (N=326,324) | 15 | 12
  Any SAEs (N=326,324) | 8 | 11
  Deaths (N=326,324) | 0 | 0
  Medically attended AEs (N=326,324) | 110 | 113
  AEs resulting in premature withdrawal (N=326,324) | 1 | 0
  AEs of Special Interest (N=326,324) | 0 | 0
  New Onset of Chronic Disease(N=326,324) | 0 | 3

10. Secondary Outcome: Geometric Mean Ratios Against A/H5N1 Strain Following 2-Dose Vaccination Schedule Of Either Low Dose Or High Dose AH5N1c Vaccine in Subjects Aged 6 to <36 Months.
Description: Immunogenicity was measured as the geometric mean ratio (GMR). The ratio of postvaccination to prevaccination HI GMTs, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination with either low dose or high dose of aH5N1c in subjects aged 6 to <36 months is reported.
  The criterion is met according to the European Committee for Medicinal Products for Human Use (CHMP) criteria if the geometric mean increase GMR (day 43/day 1) in HI antibody titer is >2.5.
  As no CHMP criteria are established for the pediatric population, criteria given for subjects 18-60 years of age were applied.
Time Frame: Day 1, day 22, day 43 and day 387
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 84 | 86
Ratio
  A/H5N1 (Day22/Day1) | 12 [7.28 to 19] | 4.56 [2.78 to 7.47]
  A/H5N1 (Day43/Day1; N=84,85) | 302 [192 to 476] | 116 [74 to 181]
  A/H5N1 (Day387/Day1; N=78,77) | 52 [25 to 106] | 19 [9.3 to 37]

11. Secondary Outcome: Geometric Mean Ratios Against A/H5N1 Strain Following 2-Dose Vaccination Schedule Of Either Low Dose Or High Dose AH5N1c Vaccine in Subjects Aged 3 to <9 Years.
Description: Immunogenicity was measured as geometric mean ratio (GMR). The ratio of postvaccination to prevaccination HI GMTs, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination with either low dose or high dose of aH5N1c in subjects aged 3 to <9 years is reported.
  As no CHMP criteria are established for the pediatric population, criteria given for subjects 18-60 years of age were applied.
  The criterion is met according to the European Committee for Medicinal Products for Human Use (CHMP) criteria if the geometric mean increase GMR (day 43/day 1) in HI antibody titer is >2.5.
Time Frame: Day 1, day 22, day 43 and day 387
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 95 | 98
Ratio
  A/H5N1 (Day22/Day1) | 9.81 [5.96 to 16] | 8.22 [4.84 to 14]
  A/H5N1 (Day43/Day1; N=93,98) | 249 [153 to 404] | 73 [44 to 121]
  A/H5N1 (Day387/Day1; N=89,94) | 11 [7.32 to 18] | 4.62 [2.92 to 7.31]

12. Secondary Outcome: Geometric Mean Ratios Against A/H5N1 Strain Following 2-Dose Vaccination Schedule Of Either Low Dose Or High Dose AH5N1c Vaccine in Subjects Aged 9 to <18 Years.
Description: Immunogenicity was measured as the geometric mean ratio (GMR). The ratio of postvaccination to prevaccination HI GMTs, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination with either low dose or high dose of aH5N1c in subjects aged 9 to <18 years is reported.
  As no CHMP criteria are established for the pediatric population, criteria given for subjects 18-60 years of age were applied.
  The criterion is met according to the European Committee for Medicinal Products for Human Use (CHMP) criteria if the geometric mean increase GMR (day 43/day 1) in HI antibody titer is >2.5.
Time Frame: Day 1, day 22, day 43 and day 387
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 102 | 105
Ratio
  A/H5N1 (Day22/Day1; N=102,103) | 15 [8.78 to 27] | 6.74 [3.93 to 12]
  A/H5N1 (Day43/Day1) | 186 [105 to 328] | 58 [34 to 101]
  A/H5N1 (Day387/Day1; N=97,100) | 4.05 [2.76 to 5.94] | 2.64 [1.83 to 3.81]

13. Secondary Outcome: Percentages Of Subjects Aged 6 to <36 Months, With HI Titers ≥40 Against A/H5N1 Strain
Description: Immunogenicity was assessed in terms of percentage of subjects aged 6 to <36 months, achieving HI titers ≥40, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination of either low dose or high dose of aH5N1c according to the CHMP criterion.
  European Licensure (CHMP) criterion is met if the percentage of subjects achieving (at day 43) HI titers ≥40 is >70%.
Time Frame: Day 1, day 22, day 43 and day 387.
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 93 | 90
Percentages of subjects
  Day 1 | 1 [0.027 to 6] | 0 [0 to 4]
  Day 22 (N=85,86) | 58 [46 to 68] | 36 [26 to 47]
  Day 43 (N=91,85) | 98 [92 to 100] | 94 [87 to 98]
  Day 387 (N=84,77) | 71 [61 to 81] | 61 [49 to 72]

14. Secondary Outcome: Percentages Of Subjects Aged 3 to <9 Years, With HI Titers ≥40 Against A/H5N1 Strain
Description: Immunogenicity was assessed in terms of percentage of subjects aged 3 to <9 years, achieving HI titers ≥40, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination of either low dose or high dose of aH5N1c according to the CHMP criterion.
  European Licensure (CHMP) criterion is met if the percentage of subjects achieving (at day 43) HI titers ≥40 is >70%.
Time Frame: Day 1, day 22, day 43 and day 387.
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 98 | 101
Percentages of subjects
  Day 1 | 0 [0 to 4] | 0 [0 to 4]
  Day 22 (N=96,98) | 43 [33 to 53] | 41 [31 to 51]
  Day 43 (N=94,98) | 98 [93 to 100] | 86 [77 to 92]
  Day 387 (90,94) | 44 [34 to 55] | 22 [14 to 32]

15. Secondary Outcome: Percentages Of Subjects Aged 9 to <18 Years, With HI Titers ≥40 Against A/H5N1 Strain
Description: Immunogenicity was assessed in terms of percentage of subjects aged 9 to <18 years, achieving HI titers ≥40, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination of either low dose or high dose of aH5N1c according to the CHMP criterion.
  European Licensure (CHMP) criterion is met if the percentage of subjects achieving (at day 43) HI titers ≥40 is >70%.
Time Frame: Day 1, day 22, day 43 and day 387.
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 103 | 109
Percentages of subjects
  Day 1 | 2 [0 to 7] | 1 [0.023 to 5]
  Day 22 (N=102,103) | 54 [44 to 64] | 37 [28 to 47]
  Day 43 (N=102,105) | 92 [85 to 97] | 79 [70 to 86]
  Day 387 (N=97,100) | 29 [20 to 39] | 17 [10 to 26]

16. Secondary Outcome: The Percentages Of Subjects Aged 6 to <36 Months, Achieving Seroconversion Against A/H5N1 Strain
Description: Immunogenicity was assessed in terms of percentages of subjects aged 6 to <36 months achieving seroconversion in HI titers, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination of either low dose or high dose aH5N1c vaccine according to the CHMP criterion.
  Seroconversion is defined as the percentages of subjects with a prevaccination HI titer <10, a postvaccination titer ≥40; or in subjects with prevaccination HI titer ≥10, and a minimum four-fold rise in postvaccination HI antibody titer.
  The criterion is met according to the European (CHMP) guideline if the percentage of subjects achieving seroconversion (at day 43) is >40%.
Time Frame: Day 22, day 43 and day 387
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 84 | 86
Percentages of subjects
  Day 22 | 58 [47 to 69] | 36 [26 to 47]
  Day 43 (N=84,85) | 99 [94 to 100] | 94 [87 to 98]
  Day 387 (N=78,77) | 73 [62 to 82] | 61 [49 to 72]

17. Secondary Outcome: The Percentages Of Subjects Aged 3 to <9 Years, Achieving Seroconversion Against A/H5N1 Strain
Description: Immunogenicity was assessed in terms of percentages of subjects aged 3 to <9 years achieving seroconversion in HI titers, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination of either low dose or high dose aH5N1c vaccine according to the CHMP criterion.
  Seroconversion is defined as the percentages of subjects with a prevaccination HI titer <10, a postvaccination titer ≥40; or in subjects with prevaccination HI titer ≥10, and a minimum four-fold rise in postvaccination HI antibody titer.
  The criterion is met according to the European (CHMP) guideline if the percentage of subjects achieving seroconversion (at day 43) is >40%.
Time Frame: Day 22, day 43 and day 387
Population: Analysis was done on FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 95 | 98
Percentages of subjects
  Day 22 | 43 [33 to 54] | 41 [31 to 51]
  Day 43 (N=93,98) | 98 [92 to 100] | 86 [77 to 92]
  Day 387 (N=89,94) | 45 [34 to 56] | 22 [14 to 32]

18. Secondary Outcome: The Percentages Of Subjects Aged 9 to <18 Years, Achieving Seroconversion Against A/H5N1 Strain
Description: Immunogenicity was assessed in terms of percentages of subjects aged 9 to <18 years achieving seroconversion in HI titers, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination of either low dose or high dose aH5N1c vaccine according to the CHMP criterion.
  Seroconversion is defined as the percentages of subjects with a prevaccination HI titer <10, a postvaccination titer ≥40; or in subjects with prevaccination HI titer ≥10, and a minimum four-fold rise in postvaccination HI antibody titer.
  The criterion is met according to the European (CHMP) guideline if the percentage of subjects achieving seroconversion (at day 43) is >40%.
Time Frame: Day 22, day 43 and day 387
Population: Analysis was done the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 102 | 105
Percentages of subjects
  Day 22 (N=102,103) | 54 [44 to 64] | 36 [27 to 46]
  Day 43 | 92 [85 to 97] | 79 [70 to 86]
  Day 387 (N=97,100) | 29 [20 to 39] | 16 [9 to 25]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events from day 1 to 7. Unsolicited AEs (other than SAEs) from day 1 to 387.
Description: All Solicited AEs are classified as systematic assessment and all unsolicited AEs are classified as non-systematic assessment.
  In total 658 subjects, who were exposed to at least one study vaccination were considered for the safety evaluation and included in overall safety set
Groups:
- Total: Total of subjects in both high dose and low dose groups.
Arm/Group | High Dose | Low Dose | Total
Serious Adverse Events (participants affected / at risk) | 8/329 | 11/329 | 19/658
Other Adverse Events (participants affected / at risk) | 263/329 | 257/329 | 520/658
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=329) | Low Dose (N=329) | Total (N=658)
FOOD POISONING (Gastrointestinal disorders) | 1 | 1 | 2
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1 | 1
CELLULITIS ORBITAL (Infections and infestations) | 1 | 0 | 1
DENGUE FEVER (Infections and infestations) | 1 | 1 | 2
GASTROENTERITIS (Infections and infestations) | 2 | 1 | 3
INFLUENZA (Infections and infestations) | 0 | 1 | 1
PNEUMONIA (Infections and infestations) | 2 | 0 | 2
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 | 1 | 1
STREPTOCOCCAL SEPSIS (Infections and infestations) | 1 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
CONVULSION (Nervous system disorders) | 0 | 1 | 1
FEBRILE CONVULSION (Nervous system disorders) | 1 | 0 | 1
APNOEIC ATTACK (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=329) | Low Dose (N=329) | Total (N=658)
NAUSEA (Gastrointestinal disorders) | 25 | 29 | 54
FATIGUE (General disorders) | 44 | 50 | 94
INJECTION SITE ERYTHEMA (General disorders) | 60 | 54 | 114
INJECTION SITE HAEMORRHAGE (General disorders) | 23 | 19 | 42
INJECTION SITE INDURATION (General disorders) | 45 | 39 | 84
INJECTION SITE PAIN (General disorders) | 209 | 213 | 422
MALAISE (General disorders) | 40 | 38 | 78
PYREXIA (General disorders) | 48 | 32 | 80
NASOPHARYNGITIS (Infections and infestations) | 18 | 16 | 34
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 55 | 58 | 113
DECREASED APPETITE (Metabolism and nutrition disorders) | 22 | 21 | 43
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 23 | 20 | 43
MYALGIA (Musculoskeletal and connective tissue disorders) | 50 | 45 | 95
HEADACHE (Nervous system disorders) | 40 | 48 | 88
SOMNOLENCE (Nervous system disorders) | 42 | 41 | 83
EATING DISORDER (Psychiatric disorders) | 29 | 20 | 49
IRRITABILITY (Psychiatric disorders) | 49 | 47 | 96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No